CLINICAL TRIAL: NCT06414993
Title: Leveraging Parents and Peer Recovery Supports to Increase Recovery Capital in Emerging Adults With Polysubstance Use: Feasibility, Acceptability, and Scaling up of Launch
Brief Title: Leveraging Parents and Peers to Increase Recovery Capital in Emerging Adults
Acronym: Launch
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chestnut Health Systems (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Tess Drazdowski, Principal Investigator, Chestnut Health Systems
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R34DA057639 (NIH); R34DA057639 (NIH)
Record Dates: First submitted 2024-05-07; First posted 2024-05-16 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Polysubstance Drug Use (Indiscriminate Drug Use)
Keywords: Contingency management; Emerging adults; Polysubstance use; Peer recovery support services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Contingency Management for Emerging Adults (CM-EA) Only (Experimental): The parents in this group will receive CM-EA delivered virtually by a parent coach approximately weekly (20-40 minute sessions) for 6 months.
  Interventions: Behavioral: Contingency Management for Emerging Adults (CM-EA)
- Standard Peer Recovery Support Services (PRSS)+Vocational/Educational (V/E) Skill Building (Experimental): The EAs in this group will receive PRSS+Vocational/Educational (V/E) Skill Building delivered by peer workers in-person in the local community and/or virtually, for approximately weekly (1 hour sessions) for 6 months.
  Interventions: Behavioral: Standard Peer Recovery Support Services (PRSS) +Vocational/Educational (V/E) Skill Building services
- CM-EA and PRSS+V/E (Experimental): Families receive both CM-EA and PRSS + V/E as described above.
  Interventions: Behavioral: Contingency Management for Emerging Adults (CM-EA); Behavioral: Standard Peer Recovery Support Services (PRSS) +Vocational/Educational (V/E) Skill Building services

INTERVENTIONS:
Behavioral: Contingency Management for Emerging Adults (CM-EA) — After CM-EA is introduced, a contingency contract is developed between a parent and emerging adult (EA) that provides EAs with rewards for negative drug screens and completion of developmentally appropriate goals to build recovery capital, along with disincentives for positive screens or engaging in inappropriate behaviors. Concurrently, parents are taught to conduct random urine drug screens. Additionally, parents are trained to complete functional analyses in collaboration with their EA to identify the EA's triggers for poly-substance use and negative behaviors. Individualized triggers are targeted via self-management planning and drug refusal skills training. At the end of CM-EA, plans are made with the family for sustaining abstinence and improvements in other behaviors.
  Arms: CM-EA and PRSS+V/E; Contingency Management for Emerging Adults (CM-EA) Only
Behavioral: Standard Peer Recovery Support Services (PRSS) +Vocational/Educational (V/E) Skill Building services — Standard PRSS begin by identifying clients' needs in key domains (e.g., transportation, employment). After needs are identified, a peer worker addresses needs through informational resources and community referrals and engages clients in positive recreational activities offering advice, hope and empowerment to encourage steps toward a reduction in substance use and eventual abstinence. When desired, peer workers also link clients to a broader recovery peer community. In addition, the peer worker will dedicate time to increasing recovery capital via improving skills related to V/E advancement using a workbook, Targeting Employment for Emerging Adults: A Toolkit for Mental Health Providers, for which peer workers will be trained.
  Arms: CM-EA and PRSS+V/E; Standard Peer Recovery Support Services (PRSS)+Vocational/Educational (V/E) Skill Building

SUMMARY:
Emerging adults (EAs; aged 18-26) are the highest-risk population for poly-substance use (misuse of more than one drug), compared to all other age groups and are the least-served population for substance use services. The overarching purpose of this pilot study is to assess whether an innovative services package, Launch, can reasonably work (is feasible) and whether providers and participants like it (acceptability). Launch works with both EAs and a supportive parent (or parental figure) and delivers peer recovery support services (PRSS) to EAs while helping parents use an effective, evidence-based program called contingency management, adapted for EAs, at home with their EA child. This study will also lay the groundwork for a future large-scale trial of Launch services.

DETAILED DESCRIPTION:
The objective of the study is to investigate a scalable service that can be used in rural communities called Launch. Launch is an innovative adaptation of current evidence-based services for Emerging Adults (EAs), ages 18-26 years old with polysubstance use (poly-SU); with a particular emphasis on increasing their recovery capital. Recovery capital is the resources available to promote substance use recovery (e.g., vocational/educational skills, recovery-supportive community). Launch leverages (1) parents of EAs and (2) peer recovery support services (PRSS), while ensuring services are equitable and scalable by using digital technology and existing substance use services infrastructure. Participants will be 48 families that include an EA struggling with poly-SU and a parent or parental figure supportive of their EA child's recovery journey. Families will be randomized to one of three conditions detailed further in the attached materials that include either: (1) Virtual Parent Contingency Management for Emerging Adults (CM-EA) Coach for parents only, (2) In-Person and/or Virtual PRSS for EAs only, or (3) a combination of Virtual Parent CM-EA Coach for parents and In-Person and/or Virtual PRSS for EAs. Quantitative and qualitative measures will assess the feasibility and acceptability of Launch. Additionally, payors/providers of substance use services will be interviewed in this study with the aim of improving future uptake and implementation of the service should it be deemed effective.

The aims of the study are as follows:

1. Adapt and evaluate the Launch parent coach and PRSS training protocols/adherence tools.
2. Assess the feasibility and acceptability of (a) a virtual study protocol for recruiting, assessing, and retaining parents and EAs and (b) Launch components.
3. Determine from payors and providers the data needed for future funding and delivery of Launch, as well as develop a site recruitment pool for a rigorous R01 trial.

ELIGIBILITY:
This study has four different participants: (1) Emerging Adult (EA)/Parent Pairs, (2) Peer Workers, (3) Parent Coaches, and (4) Payors/Providers of Recovery Services.

1. Emerging Adult (EA)/Parent Pairs

   Inclusion Criteria:
   * EA (aged 18-26) who reports (1) misuse of opioids and/or stimulants and at least one other substance in the same week during the past year, (2) at least one SU disorder reported by EA or parent as assessed via the DSM-V Checklist, and (3) has a supportive parent willing to be virtually coached to deliver CM-EA. Participating "parents" can include any supportive adult who is in a financially supportive caregiving role for the EA and has the desire and ability to implement the CM-EA program

   Exclusion Criteria:
   * Only EAs that present with unstable conditions requiring intensive treatment, such as hospital interventions, will be excluded from the sample. Examples of these conditions include participant reports of active suicidal or homicidal intentions or requests for medically supervised detox services.
2. Peer Workers

   Inclusion Criteria:
   * Certified peer worker (aged 18+) willing to be trained in vocational/educational skill building and participate in research protocols with study-enrolled emerging adult clients.

   Exclusion Criteria:
   * None
3. Parent Coaches

   Inclusion Criteria:
   * Individual (18+) with a background in clinical work willing to be trained in Contingency Management for Emerging Adults (CM-EA) and participate in research protocols with study-enrolled parent clients.

   Exclusion Criteria:
   * None
4. .Payors/Providers of Recovery Services

Inclusion Criteria:

* Individual (18+) who works at an administrative level at an organization that provides or pays for recovery services that would potentially fund or otherwise support the implementation of Launch services willing to be interviewed.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Levels of Emerging Adult Perceptions of Acceptability of the Launch Intervention (measured at 6 months). | 6 months
  Levels of acceptability of the Launch intervention, such as if participants like the intervention, as reported by emerging adults on the Acceptability of Intervention Measure. Scores range from 4-20. Higher scores indicate higher levels of intervention acceptability.
Levels of Parent Perceptions of Acceptability of the Launch Intervention (measured at 6 months). | 6 months
  Levels of acceptability of the Launch intervention, such as if participants like the intervention, as reported by parents on the Acceptability of Intervention Measure. Scores range from 4-20. Higher scores indicate higher levels of intervention acceptability.
Levels of Emerging Adult Perceptions of Launch Intervention Appropriateness (measured 6 months). | 6 months
  Levels of Launch intervention appropriateness, such as if the intervention is a good match, as reported by emerging adults on the Intervention Appropriateness Measure. Scores range from 4-20. Higher scores indicate higher levels of intervention appropriateness.
Levels of Parent Perceptions of Launch Intervention Appropriateness (measured 6 months). | 6 months
  Levels of Launch intervention appropriateness, such as if the intervention is a good match, as reported by parents on the Intervention Appropriateness Measure. Scores range from 4-20. Higher scores indicate higher levels of intervention appropriateness.
Levels of Emerging Adult Perceptions of Feasibility of the Launch Intervention (measured at 6 months). | 6 months
  Levels of Launch intervention feasibility, such as if the intervention is easy to use, as reported by emerging adults on the Feasibility of Intervention Measure. Scores range from 4-20. Higher scores indicate higher levels of intervention feasibility.
Levels of Parent Perceptions of Feasibility of the Launch Intervention (measured at 6 months). | 6 months
  Levels of Launch intervention feasibility, such as if the intervention is easy to use, as reported by parents on the Feasibility of Intervention Measure. Scores range from 4-20. Higher scores indicate higher levels of intervention feasibility.
Levels of Emerging Adult Client Satisfaction with Launch Services (measured at 6 months). | 6 months
  Levels of satisfaction with the Launch services reported by emerging adult clients on the Client Satisfaction Questionnaire 8-item scale adapted to reflect receipt of Launch services.
Levels of Parent Client Satisfaction with Launch Services (measured at 6 months). | 6 months
  Levels of satisfaction with the Launch services reported by parent clients on the Client Satisfaction Questionnaire 8-item scale (CSQ-8) adapted to reflect receipt of Launch services.

SECONDARY OUTCOMES:
Changes from baseline to 6 months post-baseline in Emerging Adult Substance Use Disorders (measured at 0 and 6 months). | Baseline to 6 months
  Frequency of substance use disorders reported by emerging adults on the Diagnostic and Statistical Manual of Mental Illnesses Version 5 (DSM-5) Substance Use Checklist for the following substance categories: alcohol, cannabis, hallucinogens, inhalants, opioids, sedatives/hypnotics/anxiolytics, stimulants, and an "other" category.
Changes from baseline to 6 months post-baseline in Emerging Adult Substance Use and Problems (measured at 0 and 6 months). | Baseline to 6 months
  Frequency of substance use and substance-related problems reported by emerging adults on the Global Appraisal of Individual Needs (GAIN) and (Justice Community Opioid Innovation Network (JCOIN) Core Measures for the past 30 days.
Changes from baseline to 6 months post-baseline in Emerging Adult Polysubstance Use (measured at 0 and 6 months). | Baseline to 6 months
  Frequency of polysubstance use reported by emerging adults on the Polysubstance Use Assessment Tool.
Changes from baseline to 6 months post-baseline in Emerging Adult Quality of Life (measured at 0 and 6 months). | Baseline to 6 months
  Levels of quality of life reported by emerging adults on the Patient-Reported Outcomes Measurement Information System (PROMIS)-29+2 Profile V2.1, a 31-item measure of quality of life across 7 domains: physical function, anxiety, depression, fatigue, sleep disturbance, social participation, pain interference, pain intensity, and cognitive function.
Changes from baseline to 6 months post-baseline in Emerging Adult Service Utilization (measured at 0 and 6 months). | Baseline to 6 months
  Frequency of service utilization in the past 30 days reported by emerging adults on the JCOIN Core Measures Service Utilization Scale, higher score indicate more service utilization.
Changes from baseline to 6 months post-baseline in Emerging Adult Abstinence Self Efficacy (measured at 0 and 6 months). | Baseline to 6 months
  Levels of abstinence self-efficacy reported by emerging adults on the Abstinence Self Efficacy Scale, higher scores indicate higher abstinence self efficacy.
Changes from baseline to 6 months post-baseline in Emerging Adult Recovery Capital (measured at 0 and 6 months). | Baseline to 6 months
  Levels of recovery capital as reported by emerging adult clients on the Emerging Adult Recovery Capital Scale, an emerging adult-specific measure under development by members of the study team and collaborators, higher scores indicate higher recovery capital.
Changes from baseline to 6 months post-baseline in Recovery Capital (measured at 0 and 6 months). | Baseline to 6 months
  Levels of recovery capital as reported by emerging adult clients on the Brief Assessment of Recovery Capital (BARC-10); higher scores indicate higher levels of recovery capital.
Levels of Emerging Adult Client Quality of Relationship with Peer Worker (measured at 6 months). | 6 months
  Levels of the quality of the relationship between the emerging adult client and the peer worker as reported by emerging adults on the Dual Role Relationship Inventory adapted to assess emerging adults' perceptions of their relationship with their peer worker (among emerging adults assigned to work with a peer worker).
Levels of Emerging Adult Client Quality of Relationship with Parent (measured at 0 and 6 months). | Baseline to 6 months
  Levels of the quality of the relationship between the emerging adult client and their parent as reported by emerging adults on the Dual Role Relationship Inventory adapted to assess emerging adults' perceptions of their relationship with their parent.
Levels of Emerging Adult Session Attendance with Peer Worker (measured weekly from baseline to 6 months). | Duration of services until 6 months after baseline
  Frequency of emerging adult attendance at their peer worker sessions (e.g., attended, no show, rescheduled) as reported by the peer worker.
Levels of Parent Session Attendance with CM-EA Parent Coach (measured weekly from baseline to 6 months). | Duration of services until 6 months after baseline
  Frequency of parent attendance at their CM-EA parent coach sessions (e.g., attended, no show, rescheduled) as reported by the parent coach.
Attitudes at 6 months post-baseline in Emerging Adult Attitudes Toward the Services Provided, Research Protocol, and Parent/Emerging Adult Relationship (measured at 6 months). | 6 months
  Emerging adult attitudes toward the Launch services program, including their perceptions of the acceptability, appropriateness, and feasibility of Launch as well as the research protocol, and impact of services on themselves and their relationship with their parents as measured during qualitative interviews with emerging adults.
Attitudes at 6 months post-baseline in Parent Attitudes Toward the Services Provided, Research Protocol, and Parent/Emerging Adult Relationship (measured at 6 months). | 6 months
  Parent attitudes toward the Launch services program, including their perceptions of the acceptability, appropriateness, and feasibility of Launch as well as the research protocol, and impact of services on their emerging adult child and their relationship with their emerging adult child as measured during qualitative interviews with parents.
Attitudes at end of services in Peer Worker Attitudes Toward the Services Provided, Impacts on Emerging Adult Clients, and Services Improvement (measured at 6 months). | From date of consent until the date of two months past last client session completed, assessed up to 2 years
  Peer worker attitudes toward the Launch services program, including their perceptions of the acceptability, appropriateness, and feasibility of Launch, the impact of services on their emerging adult clients, and suggestions for services improvement as measured during qualitative interviews with peer workers.
Attitudes at end of services in Parent Coach Attitudes Toward the Services Provided, Impacts on Parent Clients, and Services Improvement (measured at 6 months). | From date of consent until the date of two months past last client session completed, assessed up to 2 years
  Parent coach attitudes toward the Launch services program, including their perceptions of the acceptability, appropriateness, and feasibility of Launch, the impact of services on their parent clients, and suggestions for services improvement as measured during qualitative interviews with parent coaches.
Changes from baseline to end fo services in Peer Worker Services and Vocational/Educational Activity Completion (measured monthly throughout services duration). | Duration of services, after each session with an emerging adult until 6 months after baseline
  Frequency of peer worker completion of vocational/educational coaching activities reported by peer workers coaches on the Session Checklist and session tape coding.
Changes from baseline to end fo services in Parent Contingency Management for Emerging Adults (CM-EA) Adherence (measured monthly throughout services duration). | Duration of services, after each session with a parent until 6 months after baseline
  Adherence to CM-EA practices by parents reported by parent coaches as measured using the CM-Therapist Adherence Measure (CM-TAM) (Self-report version and Tape Coding version).
Descriptions of Economic-Related Information for Future Large-Scale Study from Payors/Providers of Recovery Services (measured once at any point during the study period). | Up to 2 years
  Payors and providers of recovery services will report via qualitative interviews on what kinds of participant-level outcomes or economic-related information they would want to know about as the result of a future large-scale study, selection of appropriate comparators for the future cost-effectiveness analysis, and potential recruitment sites for a future large-scale study of Launch.

CONTACTS AND LOCATIONS:
Overall Officials: Tess K Drazdowski, PhD, Principal Investigator — Chestnut Health Systems
Locations (8):
- United States (8):
  - Rising Sun Recovery, Hiram, Georgia
  - A New Horizon, Bloomington, Illinois
  - Chestnut Health Systems, Granite City, Illinois
  - Take Action Today, West Frankfort, Illinois
  - Wabash Valley Recovery Center, Terre Haute, Indiana
  - Chestnut Health Systems, Hillsboro, Missouri
  - Chestnut Health Systems, Eugene, Oregon
  - WeCare Hawkins, Rogersville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Attendance data, client satisfaction data, and EA outcomes data will be shared. Participants will be assigned a unique identifier to allow linking across data files.
  These data will be stored in an electronic file format (e.g., csv), accessible to standard analytic software (e.g., Excel, SAS) and will undergo formatting and quality assurances prior to sharing. Data dictionaries and codebooks, detailing variable-level information also will be shared.
  The PI agrees to deposit and maintain the data, and any secondary analysis of data prior to depositing data into the NAHDAP or similar repository. The PI understands that NAHDAP and similar repositories have data access policies and procedures consistent with NIH and the Helping End Addiction Long-term (HEAL) Initiative data sharing policies. HEAL data stewards will ensure that data are available to the HEAL Ecosystem after deposit.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be shared upon acceptance of the data for publication or within six months after the completion of the 6-month follow-up assessments, whichever is earlier.
Access Criteria: Information on where the data will be available and how to access the data will be included in any publications and presentations that the study team authors using these data. The repositories (e.g., NAHDAP), HEAL Data Ecosystem, and funding sources will be acknowledged in any publications and presentations. Repositories such as the NAHDAP have policies and procedures in place that will provide data access to qualified researchers, fully consistent with NIH data sharing policies and applicable laws and regulations.

REFERENCES:
- [Derived] Drazdowski TK, Castedo de Martell S, Sheidow AJ, Chapman JE, McCart MR. Leveraging Parents and Peer Recovery Supports to Increase Recovery Capital in Emerging Adults With Polysubstance Use: Protocol for a Feasibility, Acceptability, and Appropriateness Study of Launch. JMIR Res Protoc. 2024 Jul 22;13:e60671. doi: 10.2196/60671. PMID 39037768